CLINICAL TRIAL: NCT02236377
Title: Exposure, Relaxation, Rescripting Therapy (ERRT) Dismantling
Brief Title: Dismantling Exposure, Relaxation, and Rescripting Therapy
Acronym: ERRT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tulsa (Other)
Responsible Party: Principal Investigator, Joanne Davis, Associate Professor, University of Tulsa
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TU1458R1
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Frequent Trauma-related Nightmares
Keywords: ERRT; Nightmares; Sleep; Trauma; PTSD
MeSH Terms: conditions — Wounds and Injuries; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- ERRT - Enhanced Exposure (Active Comparator): Exposure, Relaxation, and Rescripting Therapy, 5 sessions, with enhanced exposure techniques
  Interventions: Behavioral: Exposure, Relaxation, and Rescripting Therapy
- ERRT - Sleep and Relaxation (Active Comparator): Exposure, Relaxation, and Rescripting Therapy protocol, 5 sessions, focused on sleep and relaxation
  Interventions: Behavioral: Exposure, Relaxation, and Rescripting Therapy
- ERRT-Rescription (Active Comparator): Exposure, Relaxation, and Rescripting Therapy, 5 sessions, with rescription but no exposure
  Interventions: Behavioral: Exposure, Relaxation, and Rescripting Therapy
- ERRT-Sleep (Active Comparator): Exposure, Relaxation, and Rescripting Therapy, 5 sessions, with enhanced sleep techniques
  Interventions: Behavioral: Exposure, Relaxation, and Rescripting Therapy
- ERRT - Consensus Manual (Active Comparator): Consensus Protocol, 6 sessions, includes components of ERRT and other nightmare protocols.
  Interventions: Behavioral: Exposure, Relaxation, and Rescripting Therapy

INTERVENTIONS:
Behavioral: Exposure, Relaxation, and Rescripting Therapy — Brief cognitive behavioral treatment targeting trauma-related nightmares and sleep problems
  Other Names: ERRT

SUMMARY:
The purpose of this case series dismantling study is to extend previous findings regarding the efficacy of a brief treatment for chronic post-trauma nightmares by examining the dose effect and mechanism of change.

Exposure, relaxation, and rescripting therapy (ERRT) is a promising psychological intervention developed to target trauma-related nightmares and sleep disturbances. ERRT has exhibited strong support in reducing the frequency and intensity of nightmares, as well as improving overall sleep quality in both civilian and veteran samples. In addition, significant decreases in PTSD and depression symptoms have been reported following treatment (Davis et al., 2011; Davis & Wright, 2007; Long et al., 2011; Swanson, Favorite, Horin, & Arnedt, 2009). ERRT is currently an evidence-level B suggested treatment (Cranston, Davis, Rhudy, & Favorite, 2011).

Despite this evidence, the mechanism of change for ERRT remains unclear. We propose to conduct a set of case series in order to examine the possible mechanisms: psycho-education, dose response for exposure, and no exposure components of the treatment. Each part of the treatment is theorized to contribute to the improved treatment outcome and it is hypothesized that participants will benefit no matter what group they are in. All participants will receive 5 to 6 treatment sessions, conducted once per week for about 90 minutes, of a modified version of ERRT.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at the time of the intake,
* experienced a traumatic event, as defined by the Diagnostic and Statistical Manual (DSM-5),
* have approximately one nightmare each week for the past month
* be able to read and speak English.

Exclusion Criteria:

* age of 17 or younger
* acute or apparent psychosis
* unmedicated bipolar disorder
* intellectual disability
* active suicidality,
* recent parasuicidal behaviors
* untreated substance use disorder in past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-08; Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Nightmare Frequency Past Week | up to 6 months followup
  This fill-in-the-blank variable assesses the number of nights the individual experienced nightmares in the past week (range = 0 - 7 nights). Higher values indicate more nights with nightmares (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Joanne L Davis, PhD, Principal Investigator — University of Tulsa
Locations (1):
- Joanne L. Davis, Tulsa, Oklahoma, United States

REFERENCES:
- [Background] Davis JL, Rhudy JL, Pruiksma KE, Byrd P, Williams AE, McCabe KM, Bartley EJ. Physiological predictors of response to exposure, relaxation, and rescripting therapy for chronic nightmares in a randomized clinical trial. J Clin Sleep Med. 2011 Dec 15;7(6):622-31. doi: 10.5664/jcsm.1466. PMID 22171201